CLINICAL TRIAL: NCT06725602
Title: Evaluation of the Arterial Occlusion Effect on Upper and Lower Limbs by the Application of Different Pre-hospital Tourniquet Models.
Brief Title: Efficacy of Prehospital Tourniquet Models for Arterial Occlusion in Upper and Lower Limbs
Acronym: TQ-BR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Roger William Freire Ronconi, PhD Researcher, University of Sao Paulo
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 79807023.9.0000.5
Record Dates: First submitted 2024-11-27; First posted 2024-12-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhage; Hypovolemic Shock; Tourniquets
Keywords: Emergency; Trauma; Hemorrhage; Tourniquets
MeSH Terms: conditions — Hemorrhage; Shock; Emergencies; Wounds and Injuries | interventions — Vagotomy, Proximal Gastric

STUDY DESIGN:
Intervention Model Description: It is a cross-sectional and self-controlled trial, aimed at collecting primary data, with randomization of the application order regarding device, laterality, segment, and blinding of the statistical analyst regarding the applied tourniquet model.
  All participants will take part in all three arms of the study (3 device models) in a randomized manner by drawing lots, so that the devices will be compared within the same participant (self-controlled). The subjects will participate on 3 non-consecutive days, during which they will draw lots to determine which device will be used, thereby distributing their participation across the three study arms in a randomized manner.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- TQ1 (CAT) (Active Comparator): Application of CAT tourniquet
  Interventions: Device: TQ - Proximal Application ("high and tight"); Device: TQ - Controlled application (2-3 inches)
- TQ2 (T-APH) (Active Comparator): Application of T-APH tourniquet
  Interventions: Device: TQ - Proximal Application ("high and tight"); Device: TQ - Controlled application (2-3 inches)
- TQ3 (SOF) (Active Comparator): Application of SOF tourniquet
  Interventions: Device: TQ - Proximal Application ("high and tight"); Device: TQ - Controlled application (2-3 inches)

INTERVENTIONS:
Device: TQ - Proximal Application ("high and tight") — Tourniquet application: proximal ("high and tight") on arms and thighs.
  Other Names: tourniquet application; proximal; "high and tight"
Device: TQ - Controlled application (2-3 inches) — TQ Application: controlled (2-3 inches proximal to the injury) on forearms and legs.
  Other Names: controlled application; 2-3 inches

SUMMARY:
The goal of this clinical trial is to compare the occlusive capability and mechanical behavior of different commercially available pre-hospital tourniquet models and the results of their application on upper and lower limbs, in order to validate the techniques proposed in international guidelines regarding proximal application on the arm and thigh ("high and tight tourniquet") and controlled application, 2 to 3 inches proximally to the injury, on the forearm and leg ("controlled tourniquet").

It is estimated that 40 volunteer individuals will be recruited, who will sign the Informed Consent Form (ICF), a group primarily composed of undergraduate and graduate students in health-related fields. Regarding inclusion and exclusion criteria, these individuals will be of both sexes, aged ≥18 and ≤60 years, with both upper and lower limbs, a Body Mass Index (BMI) ≥18.5 and ≤30 kg/m² (considering the normal and overweight range, excluding underweight and obesity ranges), and without Diabetes Mellitus (DM), Systemic Arterial Hypertension, Buerger's disease, vascular and metabolic dysfunctions affecting the limbs including lymphedema, history of neoplasms, cardiac surgeries, renal failure, recent open or closed injuries in the limbs, or any other condition suggestive of systemic or localized vascular dysfunction in the limbs.

The main questions it aims to answer are:

Null Hypothesis (H0): There are no significant differences in the occlusive capability between TQs and in the efficacy of total vascular occlusion (arteriovenous) depending on the application site among the segments (forearm, arm, leg, thigh).

Alternative Hypothesis (H1): There are significant differences in the occlusive capability between TQs and in the efficacy of total vascular occlusion (arteriovenous) depending on the application site among the segments (forearm, arm, leg, thigh).

Specific Hypothesis: TQs will present significant variations in initial tightening pressures, arterial occlusion times, and arterial occlusion pressures, evidencing differences that may affect their efficacy.

Each participant will receive a total of 8 TQ applications on the arm, forearm, leg, and thigh segments bilaterally, for each of the 3 non-consecutive collection days. Vascular occlusion will be verified using Doppler ultrasound on the radial artery for upper limbs and on the posterior tibial artery for lower limbs.

It is a cross-sectional and self-controlled trial, aimed at collecting primary data, with randomization of the application order regarding device, laterality, segment, and blinding of the statistical analyst regarding the applied tourniquet model.

DETAILED DESCRIPTION:
METHOD

It is a cross-sectional and self-controlled trial, aimed at collecting primary data, with randomization of the application order regarding tourniquet unit, laterality, segment, and blinding of the statistical analyst regarding the applied tourniquet model.

Research Ethics

The research project was approved by the Research Ethics Committee of Hospital das Clínias, Ribeirão Preto Medical School, University of São Paulo (HCFMRP/USP), in accordance with Resolution with the Certificate of Ethical Appreciation (CAAE) number 79807023.9.0000.5440.

Volunteer Recruitment and Sample

It is estimated that 40 volunteer individuals will be recruited, a group primarily composed of undergraduate and graduate students in health-related fields. The individuals will be of both sexes, aged ≥18 and ≤60 years, with both upper and lower limbs, a Body Mass Index (BMI) ≥18.5 and ≤30 kg/m² (considering the normal and overweight range, excluding underweight and obesity ranges), and without Diabetes Mellitus (DM), Systemic Arterial Hypertension, Buerger's Disease, vascular and metabolic dysfunctions affecting the limbs including lymphedema, history of neoplasms, cardiac surgeries, renal failure, recent open or closed injuries in the limbs, or any other condition suggestive of systemic or localized vascular dysfunction in the limbs.

Pre-Examination

The participants will be directed to a pre-examination room, which is air-conditioned to maintain a controlled temperature, where they will remain seated at rest for a minimum of 10 minutes for acclimatization. Individuals meeting the inclusion/exclusion criteria will be presented with the Informed Consent Form (ICF) by the principal investigator, emphasizing the procedures and risks involved in the experiment. Those who agree to participate will sign the ICF along with the principal investigator.

Data will be collected on demographic characteristics, including sex and age, and individual identifiers will be assigned to participants in the research project through an individual participation form.

Anthropometric data collection will include weight (body mass), using a digital body weight scale; height, measured with a portable stadiometer; and Body Mass Index (BMI), calculated using the formula BMI = P / (A²), where P is weight in kilograms (kg) and A is height in meters (m).

Examination

Participants will be directed to the examination room, which is air-conditioned to 23±1°C, monitored by a tabletop thermometer and hygrometer. Participants should wear suitable clothing for the exposure of their limbs, preferably attire similar to "physical education" or "swimwear".

A sequential data collection form will be used to track the collected data. Vital signs will be measured, including blood pressure (BP) and heart rate (HR), using an automatic digital wrist blood pressure monitor and a pulse oximeter.

After data collection and acclimatization, participants will undergo the application phase, which involves the use of tourniquets (TQ) on the limbs. The applications will be classified into two types: controlled, on distal segments (forearms and legs), and proximal, on proximal segments (arms and thighs).

Each participant, on each of the three data collection days, will randomly select the tourniquet model (TQm) to be used, choosing from three models: CAT®, T-APH®, and SOF®. Afterward, the tourniquet unit (TQu) will be randomly selected by the participant, with five units available for each model, along with the laterality of the first application (LFA), between the right and left sides. Once the TQu is selected, it will be removed from the options for the next participants until all units have been used.

The LFA refers to the side of the limb (right or left) where the first TQ application will take place on that day of data collection. After selected, the segments for application (arm, forearm, leg, thigh) will be randomly determined by draw by the participant. Then, the same procedure will be followed for the contralateral side. Thus, each participant will receive eight random applications each day.

The applications will occur in the sequence drawn by the participant, starting with the segments on the side of the LFA, followed by the contralateral side.

All drawings (of TQm, TQu, LFA, application section) will be conducted using an opaque and dark box for each. The individual will take, without looking, a ball with the identification of the item drawn.

Each TQ will be applied to the eight segments (bilaterally) for all participants on each collection day. This care aims to avoid biases related to ischemia-reperfusion events if the application is repeated on the same segment on the same day.

The perimetry of the limbs will be based on the application sites and the location of the application points on the upper and lower limbs, collected bilaterally on the evaluated segments immediately before the TQ application on each collection day. The forearm location will be identified in the proximal half of the forearm, between the elbow line and the intermediate line of the forearm; and the arm location will be identified in the area closest to the armpit where a TQ can be applied. The leg location will be identified as the proximal half of the leg, between the knee line and the intermediate line of the leg; and the thigh location will be identified in the area closest to the groin where a TQ can be applied. A measuring tape will be used to measure the circumference of the limb at the TQ application sites.

The acquisition of signals from the indirect measurement of the pressure generated by the devices will be done using a two-way PVC cuff, neonatal size, with a total length of 9cm, which will be positioned on the limb.

The digital manometer will be connected to the neonatal cuff, through which the compression force of the devices will be verified. The cuff will be inflated on a flat surface until it reaches 10mmHg on the manometer and then positioned at the TQ application site.

The TQ will be positioned with the area where the tightening system is located over the cuff. The pressure generated by the tourniquet, applied over the cuff, will be measured by the digital manometer.

The tourniquets will be applied in the phases designated here: a) Initial application - consists of, after positioning the TQ around the limb, tightening the TQ by pulling its strap and securing it according to the model (using Velcro on the CAT® and TAPH® and the buckle system on the SOF®); b) Tightening and securing - consists of using the mechanical advantage system of the devices, twisting the rods until the distal pulse ceases, followed by the final locking of the rod, according to each model; c) Maintenance and removal - consists of maintaining the TQ for 30 seconds after the pulse ceases and final locking, to verify if there is a return of arterial flow during the period, and its removal, ending the application at the site.

Doppler ultrasound will be used for spectral analysis of distal flow, quantifying arterial flow before and after the application, as well as for defining the moment of arterial occlusion (absence of pulse and flow). The radial artery and the posterior tibial artery will be used for distal pulse analysis.

To address current questions about possible differences between application sites due to controlled and proximal techniques, the variables to be evaluated are: a) Initial tightening pressure (ITP) expressed in mmHg, corresponding to the pressure the device produces in the initial application, before the rod tightening; b) Arterial occlusion (AO), indicated as positive (if it occurred) or negative (if it did not occur); c) Arterial flow (ArtF), related to the pre- and post-application periods, corresponding to the systolic peak velocity (SPV) in cm/s; d) Time to arterial occlusion (TAO), expressed in seconds, from the beginning of the application to the determination of absence of flow after locking; e) Arterial occlusion pressure (AOP), expressed in mmHg, corresponding to the pressure recorded at the determination of absence of flow after locking; and f) Index of Experienced Discomfort (IED), through an adapted questionnaire.

The collection sequence for each segment involves: a) Positioning the neonatal cuff at the application site, inflated to 10mmHg, and positioning the TQ around the limb over the cuff, without tightening; b) Locating, through ultrasound/Doppler, pulse and arterial flow in the radial and posterior tibial arteries; c) Obtaining and recording pulse and ArtF data, pre-application; d) Starting the time counting and performing the initial tightening, which involves tightening the TQ strap over the cuff; e) Obtaining and recording ITP data; f) Performing mechanical advantage tightening of the device, through the rod twisting, until the arterial flow ceases (AO); g) Locking the device according to its system, where the twisting rod is locked in a specific system for each TQm; h) Reassessing pulse and flow and, if the flow has returned, unlocking the device and re-tightening (increasing the tightening by twisting the rod), locking again and recording AO as negative if the flow cessation does not occur in two tightening attempts; i) Finalizing the time count after cessation and locking, starting a 30-second count; after the period, obtaining and recording application time data, AOP, and post-application pulse and arterial flow data, if the flow cessation was maintained; if the occlusion was not maintained, recording AO as negative after the 30-second period; j) Obtaining discomfort data through the IED.

The IED will be used to evaluate the period between the device's locking and the 30-second maintenance period. It involves using the Visual Analog Scale (VAS), related to classic studies that grade uncomfortable sensations and pain from "absent" to "the worst possible", in association with the Wong-Baker Faces Pain Scale (WBFS), adapted to classify discomfort. The scale will include six images, associated with a digital visual scale with digits from 0 to 10, ranging from "no pain" to "maximum pain."

In this study, its association with the visual scale was included to better illustrate the discomfort scale and allow for better interpretation by the experiment's volunteers.

A checklist of experienced and reported discomforts or symptoms will be included, allowing for the selection of more than one option, using the terms and possibilities: "none," "pain," "decreased sensitivity," "total loss of sensitivity," "tingling," "shock sensation," "burning sensation," "I don't know how to explain," and "other," to be described.

Data Analysis

The data will undergo a normality test and, in case of non-normality, will be adjusted to a ranking format. Continuous variable data will be analyzed using a three-way repeated measures analysis of variance (ANOVA), investigating main effects and interactions between groups and within groups, using the following factors:

1. LOCATION: the relationship between upper and lower limbs, at the forearm, arm, leg, and thigh segments; and
2. TOURNIQUET: the relationship between TQm.

Data analysis will follow the characteristics of a self-controlled trial, verifying the models and locations compared within the same individual.

To determine the best TQ model among the data and variables, Bonferroni's post hoc test will be used. For non-continuous variables, the Chi-squared test will be applied.

The statistical analyst will be blinded to the device model under evaluation, having only the description "TQ1," "TQ2," and "TQ3."

HYPOTHESIS

Null Hypothesis (H0) - There are no significant differences in occlusive capacity between the mTQ and in total vascular occlusion efficacy (arteriovenous) depending on the application between segments (forearm, arm, leg, thigh).

Alternative Hypothesis (H1) - There are significant differences in occlusive capacity between the mTQ and in total vascular occlusion efficacy (arteriovenous) depending on the application between segments (forearm, arm, leg, thigh).

Specific Hypothesis - The mTQ will present significant variations in initial tightening pressures, times to arterial occlusion, and arterial occlusion pressures, highlighting differences that may affect their efficacy.

RISKS AND BENEFITS

Risks - It is common for mild to moderate pain sensations and bruising to occur at the application sites due to the device pressure against the skin, even with short-duration applications as in this study. In real-life tourniquet applications, where the device is tightened and maintained for longer periods until surgical care is provided, literature shows that consequences may arise, with highly variable incidence. Although approximately 82% of cases may have no consequences, complications from device use have been reported, including rhabdomyolysis (about 13%), fasciotomy (about 10%), nerve paresis (about 5-10%), thromboembolic events (about 6-9%), pulmonary complications (about 7%), acute renal failure (about 2-4%), cardiac complications (about 3%), ischemia-reperfusion injury (about 3%), and amputation (about 0-1%).

Some of these conditions are mainly related to traumatic injuries (in cases where the device was indicated for use) and the critical conditions of the patients. In this study, with controlled applications and short durations, such manifestations are unlikely, except for the expected ones, such as pain and bruising at the application site, as well as paresthesia during the vascular occlusion period.

Benefits - This trial does not intend to treat or provide direct health benefits to the participants. Its development will allow the evaluation of the relationship between application techniques and the effectiveness of the studied devices.

EXPECTED RESULTS

This study aims to present data related to the total vascular occlusion capacity of each device, as well as the pressure they generate and the application time required to achieve it, allowing comparisons of data between TQ models and application conditions based on the location (arm, forearm, leg, thigh).

ELIGIBILITY:
Inclusion Criteria:

* have all four limbs (both upper and lower limbs)
* Body Mass Index (BMI) ≥18.5 and ≤30 kg/m² (considering the normal and overweight range, excluding underweight and obesity ranges)

Exclusion Criteria:

* Diabetes Mellitus (DM)
* Systemic Arterial Hypertension
* Buerger's Disease
* Vascular and metabolic dysfunctions affecting the limbs including lymphedema
* history of neoplasms
* history of cardiac surgeries
* history of renal failure
* recent open or closed injuries in the limbs
* any other condition suggestive of systemic or localized vascular dysfunction in the limbs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterial Occlusion (AO) | The measurements will be assessed after the volunteer has completed all 3 days of data collection, allowing for a comparison of the 3 study arms (TQ models).
  Dichotomous variable indicated as POSITIVE (if it occurred) or NEGATIVE (if it did not occur). Variable measured immediately after the Tightening and Securing phase, in each application.
Arterial Occlusion Pressure (AOP) | The measurements will be assessed after the volunteer has completed all 3 days of data collection, allowing for a comparison of the 3 study arms (TQ models).
  Continuous variable, expressed in mmHg, corresponding to the pressure exerted by the TQ on the cuff, recorded at the confirmation of arterial occlusion after locking the device. It is measured immediately after the Tightening and Securing phase, in each TQ application.

SECONDARY OUTCOMES:
Initial Tightening Pressure (ITP) | The measures will be assessed after the volunteer has participated in all 3 days of data collection, to compare the 3 arms of the study (TQ models).
  Continuous variable expressed in mmHg, which corresponds to the pressure the device produces at initial application, before tightening by twisting the rod. It is measured in each application, immediately after the "Initial application" phase, which consists of, after positioning the TQ around the limb, tightening the TQ by pulling its strap and securing it, according to the TQm (using velcro on the CAT® and TAPH® and the buckle system on the SOF®).

OTHER OUTCOMES:
Index of Experienced Discomfort (IED) | The measurements will be assessed after the volunteer has completed all 3 days of data collection, allowing for a comparison of the 3 study arms (TQ models).
  Qualitative ordinal variable, obtained through an adapted questionnaire, used to evaluate the period between the device's locking and the post 30-seconds, in each TQ application. It involves Visual Analog Scale (VAS) in association with the Wong-Baker Faces Pain Scale (WBFS), adapted to classify discomfort. The scale will include six images, associated with a digital visual scale with digits from 0 to 10. Every 2 digits, the participant identifies, alongside the Wong-Baker faces, the expressions: 'does not hurt = 0', 'hurts a little = 2', 'hurts a little more = 4', 'hurts a lot = 6', 'hurts much more = 8', and 'hurts the most = 10'. The participant is also asked to relate any symptoms they experience, including none, pain, decreased sensitivity, total loss of sensitivity, tingling, shock sensation, burning sensation, unable to explain, or any other symptom they wish to describe.
Time to arterial occlusion (TAO) | The measurements will be assessed after the volunteer has completed all 3 days of data collection, allowing for a comparison of the 3 study arms (TQ models).
  Discrete variable, expressed in seconds, measured from the start of the TQ application to the confirmation of arterial occlusion after locking.

CONTACTS AND LOCATIONS:
Overall Officials: Roger W F Ronconi, PT, MSc, PhD(c), Principal Investigator — Faculdade de Medicina de Ribeirão Preto da USP (FMRP-USP)
Locations (1):
- Ribeirão Preto Medical School USP (FMRP-USP), Experimental Surgery Department, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will not be shared as they will be used solely for the purposes of this study.